CLINICAL TRIAL: NCT03167879
Title: Integrating Counseling to Transform HIV Family Planning Services
Brief Title: Integrating Safer Conception Counseling to Transform HIV Family Planning Services
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: RAND (Other)
Collaborators: Children's Mercy Hospital Kansas City (Other); Makerere University (Other); The AIDS Support Organization (Other); University of Kansas (Other); Eunice Kennedy Shriver National Institute of Child Health and Human Development (NICHD) (NIH)
Responsible Party: Sponsor
Allocation: Randomized | Model: Factorial | Masking: None | Purpose: Prevention
Other Study IDs: 2016-0560; R01HD090981 (NIH)
Record Dates: First submitted 2017-05-23; First posted 2017-05-30 (Actual); Results first posted 2022-11-21 (Actual); Last update posted 2022-11-21 (Actual); Status verified 2022-10

CONDITIONS: Safer Conception Intervention Trial
Keywords: family planning; safer conception; HIV; serodiscordant couples; Uganda; contraception

STUDY DESIGN:
Intervention Model Description: This 3-arm cluster RCT will compare (1) a multi-component intervention that integrates safer conception counseling (SCC) into existing family planning (FP) services and provides intensive training and supervision (SCC1), (2) the integration of the same intervention as in (1) into FP services but with a less intensive training and supervision model that mimics the Ministry of Health approach, and (3) usual care FP services, at 6 HIV clinics (2 per arm) operated by TASO Uganda. The model is factorial because the two active intervention arms will be combined and compared to usual care in some analyses.
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (3):
- SCC1--high intensity supervision (Experimental): Integration of safer conception counseling into family planning services, with intensive training and supervision
  Interventions: Behavioral: safer conception counseling
- SCC2-- low intensity supervision (Experimental): Integration of safer conception counseling into family planning services, with less intensive training and supervision that mimics Ministry of Health approach
  Interventions: Behavioral: safer conception counseling
- Usual care family planning services (No Intervention): Family planning services that are currently available as part of usual care, which focus almost solely on contraception and pregnancy prevention

INTERVENTIONS:
Behavioral: safer conception counseling — Multi-component counseling to help HIV-affected couples to make an informed decision about childbearing, and to provide counseling to use contraception or safer conception methods, depending on whether the couples chooses to seek or prevent pregnancy after initial consultation.
  Other Names: SCC
  Arms: SCC1--high intensity supervision; SCC2-- low intensity supervision

SUMMARY:
This 3-arm cluster randomized controlled trial (RCT) will compare (1) a comprehensive family planning (FP) program that incorporates a structured, multi-component safer conception counseling (SCC) intervention (SCC1) versus (2) a SCC training workshop for FP nurses (SCC2; less intensive and mimics approach used by Ugandan Ministry of Health (MoH) to integrate new services), and (3) existing FP services (usual care) at 9 HIV clinics (3 per arm) operated by The AIDS Support Organization (TASO) Uganda.

DETAILED DESCRIPTION:
Family planning (FP) services for people living HIV/AIDS (PLHA) focus on preventing unplanned pregnancies and mother-to-child-transmission (PMTCT), and currently provide no services to support safer conception, despite ~40% of HIV+ women in sub-Saharan Africa (SSA) becoming pregnant post HIV diagnosis. Antiretroviral therapy (ART) greatly reduces the transmission risks associated with childbearing, but many PLHA are either not on ART or not adequately adherent; hence the need for using safer conception methods (SCM) such as manual self-insemination and timed unprotected intercourse. This cluster RCT will compare (1) a comprehensive FP program that incorporates a structured, multi-component SCC intervention (SCC1) versus (2) an SCC training workshop for FP nurses (SCC2; mimics approach used by Ugandan MoH to integrate new services), and (3) existing FP services (usual care) at 6 HIV clinics operated by TASO Uganda. The 3-arm design, together with the planned cost-effectiveness analysis, allows us to examine two models for integrating SCC into FP services that differ on level of intensity, thereby informing MoH policy and resource allocation. Sixty clients in HIV serodiscordant relationships who express childbearing desires at recruitment will be enrolled at each site (n=360) and followed for 12 months or completion of pregnancy (if applicable). The primary outcome is use of either SCM (for those trying to conceive) or dual contraception (those who decide against pregnancy).

ELIGIBILITY:
Inclusion Criteria:

1. HIV+ client of TASO
2. Client if of reproductive age (males age 15-60; females age 15-45).
3. Has a partner with whom the client is considering having a child.
4. If client or their partner is age 15-17, the couple must be "married", defined as cohabitating and the parents of the minor(s) are reported to be aware of the relationship.
5. Partner with whom the client is considering having a child is HIV-negative.

5. Client reports that their partner is aware of the client being HIV-positive.

Exclusion Criteria:

1. Female client (or partner of male client) is pregnant

Ages: 15 Years to 60 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult
Enrollment: 389 (Actual)
Dates: Start 2017-06-15 (Actual); Primary Completion 2020-05-23 (Actual); Study Completion 2020-05-23 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Glenn Wagner, PhD, Principal Investigator — RAND
Locations (1):
- TASO, Mbale, Entebbe, Jinja, Masaka, Mbarara, Runkangiri, Uganda

IPD SHARING:
Plan to Share IPD: Yes
A data sharing plan is in place to provide a de-identified dataset to researchers who request access or through an NIH-affiliated repository

REFERENCES:
- [Derived] Wagner GJ, Wanyenze RK, Beyeza-Kashesya J, Gwokyalya V, Hurley E, Mindry D, Finocchario-Kessler S, Nanfuka M, Tebeka MG, Saya U, Booth M, Ghosh-Dastidar B, Linnemayr S, Staggs VS, Goggin K. "Our Choice" improves use of safer conception methods among HIV serodiscordant couples in Uganda: a cluster randomized controlled trial evaluating two implementation approaches. Implement Sci. 2021 Apr 15;16(1):41. doi: 10.1186/s13012-021-01109-z. PMID 33858462
- [Derived] Wagner GJ, Mindry D, Hurley EA, Beyeza-Kashesya J, Gwokyalya V, Finocchario-Kessler S, Wanyenze RK, Nanfuka M, Tebeka MG, Goggin K. Reproductive intentions and corresponding use of safer conception methods and contraception among Ugandan HIV clients in serodiscordant relationships. BMC Public Health. 2021 Jan 19;21(1):156. doi: 10.1186/s12889-021-10163-7. PMID 33468072
- [Derived] Goggin K, Hurley EA, Beyeza-Kashesya J, Gwokyalya V, Finocchario-Kessler S, Birungi J, Mindry D, Wanyenze RK, Wagner GJ. Study protocol of "Our Choice": a randomized controlled trial of the integration of safer conception counseling to transform HIV family planning services in Uganda. Implement Sci. 2018 Aug 14;13(1):110. doi: 10.1186/s13012-018-0793-y. PMID 30107843

RESULTS

PARTICIPANT FLOW:
Units Other Than Participants: clinics
Period: Overall Study
Arm/Group | SCC1--high Intensity Supervision | SCC2-- Low Intensity Supervision | Usual Care Family Planning Services
Started | 129; 2 clinics | 130; 2 clinics | 130; 2 clinics
Completed | 122; 2 clinics | 125; 2 clinics | 122; 2 clinics
Not Completed | 7; 0 clinics | 5; 0 clinics | 8; 0 clinics

BASELINE CHARACTERISTICS:
Groups:
- Total: Total of all reporting groups
Arm/Group | SCC1--high Intensity Supervision | SCC2-- Low Intensity Supervision | Usual Care Family Planning Services | Total
Number analyzed (Participants) | 129 | 130 | 130 | 389
Age, Continuous [Mean (Standard Deviation); unit: years] | 35.1 (7.2) | 35.3 (8.0) | 37.1 (9.1) | 35.9 (8.2)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 78 | 66 | 51 | 195
  Male | 51 | 64 | 79 | 194
Ethnicity (NIH/OMB) [Count of Participants; unit: Participants]
  Hispanic or Latino | 0 | 0 | 0 | 0
  Not Hispanic or Latino | 129 | 130 | 130 | 389
  Unknown or Not Reported | 0 | 0 | 0 | 0
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 0 | 0 | 0 | 0
  Asian | 0 | 0 | 0 | 0
  Native Hawaiian or Other Pacific Islander | 0 | 0 | 0 | 0
  Black or African American | 129 | 130 | 130 | 389
  White | 0 | 0 | 0 | 0
  More than one race | 0 | 0 | 0 | 0
  Unknown or Not Reported | 0 | 0 | 0 | 0
Region of Enrollment [Number; unit: participants]
  Uganda | 129 | 130 | 130 | 389
Currently on ART [Count of Participants; unit: Participants] — Whether or not the participant was currently prescribed antiretroviral therapy (ART) at the time of the assessment was obtained via chart abstraction; this is a binary variable (counting those currently on ART)
  Participants
    Currently on ART | 129 | 128 | 128 | 385
    Not currently on ART | 0 | 2 | 2 | 4
Undetectable HIV viral load [Count of Participants; unit: Participants] — HIV viral load data was abstracted from clinic charts; this variable is binary and represents whether or not the participant's last viral load at the time of the assessment was undetectable (< 20 copies per cubic millimeter) or not.
  Participants
    Last viral load was undetectable | 90 | 78 | 97 | 265
    Last viral load was not undetectable | 39 | 52 | 33 | 124

OUTCOME MEASURES:

1. Primary Outcome: Number of Participants Who Used Dual Contraception or Safer Conception Method
Description: Number of participants who used either of these methods based on the choice of the client to seek childbearing or pregnancy prevention following intervention
Time Frame: Month 12
Population: The primary analyses followed an intent-to-treat (ITT) approach (i.e., outcomes with missing data are designated as not engaging in the desired behavior or achieving the desired pregnancy status); therefore, all participants were included in analysis.
Measure: Count of Participants; unit: Participants
Arm/Group | SCC1--high Intensity Supervision | SCC2-- Low Intensity Supervision | Usual Care Family Planning Services
Number analyzed (Participants) | 129 | 130 | 130
Participants | 35 | 19 | 9
Statistical Analysis 1: Comparison: SCC1--high Intensity Supervision vs SCC2-- Low Intensity Supervision vs Usual Care Family Planning Services; Test type: Superiority; Odds Ratio (OR) = 10.63, 95% CI 2-sided [2.79 to 40.49]

2. Secondary Outcome: Number Who Achieved Desired Pregnancy Status
Description: Number who achieved desired pregnancy status depending on what client chooses after safer conception consultation
Time Frame: Month 12
Population: Analysis conducted only among those trying to conceive (n=276)
Measure: Count of Participants; unit: Participants
Arm/Group | SCC1--high Intensity Supervision | SCC2-- Low Intensity Supervision | Usual Care Family Planning Services
Number analyzed (Participants) | 104 | 87 | 85
Participants | 32 | 29 | 27
Statistical Analysis 1: Comparison: SCC1--high Intensity Supervision vs SCC2-- Low Intensity Supervision vs Usual Care Family Planning Services; Test type: Superiority; Odds Ratio (OR) = 0.73, 95% CI 2-sided [0.25 to 2.09]

3. Secondary Outcome: Partner HIV Status
Description: Partner HIV status as determined by HIV antibody test conducted by study
Time Frame: study end point (Month 12 or when learning of pregnancy)
Population: The primary analyses followed an intent-to-treat (ITT) approach (i.e., outcomes with missing data are designated as having negative outome)
Measure: Count of Participants; unit: Participants
Arm/Group | SCC1--high Intensity Supervision | SCC2-- Low Intensity Supervision | Usual Care Family Planning Services
Number analyzed (Participants) | 129 | 130 | 130
Participants
  Number who tested HIV-positive | 0 | 1 | 0
  Number who tested HIV-negative | 129 | 129 | 130
Statistical Analysis 1: Comparison: SCC1--high Intensity Supervision vs SCC2-- Low Intensity Supervision vs Usual Care Family Planning Services; Test type: Superiority; Odds Ratio (OR) = 2.23, 95% CI 2-sided [0.02 to 257.6]

4. Other Pre Specified Outcome: Cost-effectiveness of Safer Conception Counseling Intervention
Description: We tracked all costs associated with implementing SCC1 and SCC2 beyond those of existing FP services, such as labor costs associated with SCC sessions and consults with FP nurses, supervision of the FP nurses (in SCC1), contraceptives and SCM client kits, and cost of intervention materials (posters, SCM instructional videos). We assessed the costs for accurate use of SCM on its own among those trying to conceive. Because supervisors in SCC1 were research staff with significantly higher salaries than the MoH supervisors in SCC2, we conducted an additional more realistic "scale-up scenario" showing the costs of SCC1 if its supervisors' salaries were the same as the MoH supervisors' salaries. The cost-effectiveness ratio was calculated as the cost per participant divided by the relative effect size in that group compared to the usual care control.
Time Frame: 30 months of intervention implementation
Population: The primary analyses followed an intent-to-treat (ITT) approach. Cost-effectiveness data were not collected for the usual care arm.
Measure: Mean (Standard Deviation); unit: US dollars
Arm/Group | SCC1--high Intensity Supervision | SCC2-- Low Intensity Supervision | Usual Care Family Planning Services
Number analyzed (Participants) | 129 | 130 | 0
US dollars | 520 (78) | 1014 (152) |

ADVERSE EVENTS:
Time Frame: 12 month study participation
Arm/Group | SCC1--high Intensity Supervision | SCC2-- Low Intensity Supervision | Usual Care Family Planning Services
All-Cause Mortality (participants affected / at risk) | 0/129 | 0/130 | 0/130
Serious Adverse Events (participants affected / at risk) | 0/129 | 0/130 | 0/130
Other Adverse Events (participants affected / at risk) | 0/129 | 0/130 | 0/130

LIMITATIONS AND CAVEATS:
No survey data were collected from the partner of the index participant, except for female partners of male participants who were briefly interviewed on contraception use. Data reported by the female partners were recorded as data for the male participant. These female partner participants are not included in the number enrolled.

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: No

DOCUMENTS (1):
  • Study Protocol and Statistical Analysis Plan (2017-05-01): https://cdn.clinicaltrials.gov/large-docs/79/NCT03167879/Prot_SAP_000.pdf